CLINICAL TRIAL: NCT01660048
Title: Prospective Randomized Single Blind Controlled Study Comparing Single and Multiport Laparoscopic Total Extraperitoneal Inguinal Hernia Repair
Brief Title: A Prospective Study Comparing Single and Multiport Laparoscopic Inguinal Hernia Repair
Acronym: SILSTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Sydney Hernia Specialists Clinic (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Principal Investigator, Dr Hanh Minh Tran, Director, The Sydney Hernia Specialists Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HTranSILStrial; Holroyd Private Hospital (Other: Holroyd Private Hospital)
Record Dates: First submitted 2012-07-31; First posted 2012-08-08 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Inguinal Hernia
Keywords: Laparoscopic total extraperitoneal Inguinal hernia repair
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SILS TEP repair (Experimental): Half of the patients will undergo laparoscopic total extraperitoneal inguinal hernia repair using a single port (Triport)
  Interventions: Procedure: SILS TEP repair; Procedure: Total extraperitoneal inguinal hernia repair
- Multiports TEP repair (Active Comparator): Half of the patients will undergo the conventional multiports total extraperitoneal inguinal hernia repair
  Interventions: Procedure: Total extraperitoneal inguinal hernia repair

INTERVENTIONS:
Procedure: SILS TEP repair — perform the laparoscopic total extraperitoneal inguinal hernia repair using a single port
  Other Names: single port inguinal hernia repair
  Arms: SILS TEP repair
Procedure: Total extraperitoneal inguinal hernia repair — Conventional multiport laparoscopic total extraperitoneal inguinal hernia repair
  Other Names: Laparoscopic TEP inguinal hernia repair

SUMMARY:
Since laparoscopic inguinal hernia was introduced in 1990, it has now become the most commonly performed hernia repair in NSW. Traditionally this is done with 3 small incisions: a 2 cm incision under the navel for insertion of the camera and two 1 cm incisions below the navel for insertion of trocars into which dissecting instruments are inserted to perform the repair. Although this method has been shown to be relatively safe and efficient there are reports of bowel and vascular injuries from the insertion of the smaller trocars which are usually sharp. These can cause serious injuries.

Since 2009, a newer method of performing the key hole repair has been developed. This involves placing a special single port under the navel via a 2-2.5cm incision and into which 3 blunt trocars are inserted. This negates the risks of injuries from sharp trocars. In addition the fact that only a single incision is used this could potentially result in less pain, reduced incidence of wound complications including infection and improved cosmetic results.

However these potential advantages have not been proven in rigorous clinical studies as the single port technique is still relatively new. It is hoped that this study will prove that the single port technique is at least as effective and efficient as the conventional technique in the cure of hernias and may have additional benefits as enumerated above.

Neither you nor your surgeon will know which procedure (three port or single port hernia repair) until you are already asleep in the operating room and a random number selecting process will automatically assign you to one procedure or the other. Sometimes it is not possible to perform the single port safely in which case your procedure will be converted to a three ports procedure.

All patients having surgical treatment of groin hernia at Holroyd Private Hospital are subject to very careful assessment and study. All patients are requested to report immediately if there are any problems. Any problems would normally be reported to your treating surgeon who has primary responsibility for your care. Problems can be reported directly to Holroyd Private Hospital. Any information in your medical records is subject to stringent confidentiality requirements. The hospital is bound by the Australian Privacy Council Charter as regards confidentiality and privacy.

DETAILED DESCRIPTION:
This study will compare the Laparoscopic TEP repair of inguinal/femoral hernias using the traditional three ports and the newer single port techniques.

Laparoscopic hernia repair was first introduced in 1990. The uptake rate was slow to start off with such that in 1994 only 9.7% of all inguinal hernias were performed laparoscopically However, in 2009, the figure now stands at 40% Australia-wide. (www.medicareaustralia.gov.au). Indeed, in NSW this figure stands at 48%, which means that it is the commonest operation performed for inguinal hernias in this State.

Up to 2009, the laparoscopic hernia repair involves the insertion of 3 ports: 10mm port in the infra-umbilical region for the camera via a 2 cm incision and 2 x 5mm working ports usually in the midline for the dissecting instruments via 2 x 10mm incisions. These ports are called secondary trocars which are usually sharp. Their insertion has the potential to cause bowel and vascular injuries.

The European Hernia Society guidelines (www.herniaweb.org) on the treatment of inguinal hernias have shown (conventional) endoscopic techniques to be associated with higher rates of port-site hernias and visceral injuries especially during the learning curve period.

A recent study of 37,000 gynaecological laparoscopies in the US showed a bowel injury rate of 0.16%; a third of these led to the death of the patients. 22% of all bowel injuries resulted from the insertion of secondary trocars (www.danaise.com/vascular_and_bowel_injuries_duri.htm).

Another report from a large hernia centre in the US showed that in the first 300 transabdominal preperitoneal (TAPP) repairs 2 bowel injuries (and one bladder injury) were observed. Indeed, when these investigators changed the technique to a TEP repair they also observed 2 bowel injuries (and one bladder injury) in the first 300 TEP repairs. (www.ncbi.nlm.nih.gov/pubmed/11178763)

Therefore bowel and vascular injuries during laparoscopic surgery are real but they are often under reported.

Single incision laparoscopic surgery, where all the instruments are placed in a single port, has the primary aim of preventing vascular and bowel injury through the use of completely blunt trocars. The first case of laparoscopic TEP repair was reported in 2009. Since then there have only been a handful of reports.

The principle author, Dr Hanh Tran, has been performing single incision laparoscopic hernia repair since October 2009. To date, he has performed in excess of 100 cases with excellent results in terms of success of the cure of hernias (no recurrence has been observed in any of these patients although the follow-up has only been up to 1 year), no complications including wound infection, high patient satisfaction and excellent cosmetic results.

However Dr Tran's experience is at best an audit. The highest level of scientific evidence regarding the efficacy and safety of one procedure versus another comes from a prospective randomised controlled study where two procedures are compared and the patients (with their informed consent) will undergo either procedure in a random (blind) fashion.

It is proposed that 100 patients will be enrolled into the study with 50 patients in each arm of the study ie 50 patients will undergo TEP repair using the conventional three ports and 50 with the single port technique.

The TEP inguinal hernia repair is exactly the same in both procedures except in the single port technique only one (1.5-2cm) infra-umbilical incision is required. While the first 100 cases were performed with the SILS (TM) port this required a relatively larger infraumbilical incision. The availability of the Triport (TM) allows an equally small if not smaller infraumbilical incision and this would be suited to all patients rather than those with a naturally large umbilicus. Over 180 TEP inguinal hernia repairs were performed with the Triport before the commencement of the trial to ensure that the learning curve has been truly passed. Therefore the use of the Triport allows for just one inconspicuous incision compared to three incisions for the conventional multiport inguinal hernia repair with possible improved cosmetic results.

The main disadvantage of the single port technique is the relative loss of triangulation and the principle author has shown that this can be overcome with the use of a longer and smaller laparoscope (of which Holroyd Private Hospital has bought two specifically for this purpose), different dissecting techniques and with increased experience. Therefore, if a surgeon is not experienced with this technique the operation and its success can be compromised by inadequate dissection. The author (who has performed nearly 2000 TEP repairs over the past 10 years) believes that the learning curve for single port TEP hernia repair for a highly experienced TEP surgeon is around 25-50 ie after this number the operation time will approach that of the standard three ports TEP repair. He has performed in excess of 100 Single Port Incision Laparoscopic hernia repairs over the past year. Therefore the success of the operation for patients in either arm of the study will not be compromised by lack of experience.

The follow up of these patients will be no different to those followed up under the protocol of the Sydney Hernia Clinic. This is a standard follow up and is consistent with normal clinical practice.

In summary, the goals are simple. (i) To perform laparoscopic TEP inguinal hernia repair using either the conventional three ports or single port technique; (ii) To assess the efficacy of the newer single port technique in a rigorous scientific manner; (iii) To report any unexpected problems or complications; (iv) To follow up patients treated laparoscopically to ensure that the single port technique has as good results as or better in terms of cure of hernia (absence of recurrence of the hernia) and less complications and better cosmetic results as that which is achieved when the traditional 3-ports technique is used.

ELIGIBILITY:
Inclusion Criteria:

* all referred patients with inguinal hernias

Exclusion Criteria:

* workers Compensation cases
* previous extraperitoneal intervention
* unfit for a general anaesthetic
* strangulated hernias
* present of or previous ventral hernia repair extending 5 cm below umbilicus

Ages: 16 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-12; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Conversion to multiport or open operation | during operation
  This refers to whether any single port procedure needs to be converted to multiports or open procedure. This is quite a normal process as a proportion of multiport procedures are converted to open procedures for safety reasons.

SECONDARY OUTCOMES:
Operating time | during operation
  This assess the time taken to perform the operation and is defined as time from initial skin incision to complete wound closure
Length of hospital stay | day procedure or overnight stay
  This assess how long patient stays in hospital whether it is a day procedure or whether they need to stay in hospital overnight or longer
Pre and post operative pain scores | preop, day one and day 7 postop
  This utilizes the visual analogue pain score 0-10 and the patients are assessed preoperatively, day 1 and day 7 after surgery
Analgesic requirements | one week
  This assesses how many painkiller tablets (Dextropropoxyphene) patients ingest in the first week after operation
return to work or normal physical activities | 6 weeks
  This assesses how soon patients return to work or normal physical activities
Quality of life health scores | preop, 6 weeks and 1 year postop
  SF36 forms are completed before operation, 6 weeks and 1 year after operation
Cosmetic scar score | 6 weeks
  patients will be asked to assess satisfaction of their own scars 6 weeks after surgery
Recurrence of hernia | 1 year
  Patients will be assessed at 1 week, 6 weeks and one year to detect presence of recurrence of hernia
post-operative complications including urinary retention, wound infection, seroma formation, chronic pain, testicular atrophy | 6 weeks
  Patients will be seen at 1 week, 6 weeks to assess for any peri-operative complications associated with hernia surgery as enumerated above

CONTACTS AND LOCATIONS:
Overall Officials: Hanh M Tran, MD, FRACS, Principal Investigator — Sydney Hernia Specialists Clinic
Locations (1):
- Holroyd Private Hospital, Guildford, New South Wales, Australia

REFERENCES:
- [Result] Tran H. Robotic single-port hernia surgery. JSLS. 2011 Jul-Sep;15(3):309-14. doi: 10.4293/108680811X13125733356198. PMID 21985715
- [Result] Tran H. Safety and efficacy of single incision laparoscopic surgery for total extraperitoneal inguinal hernia repair. JSLS. 2011 Jan-Mar;15(1):47-52. doi: 10.4293/108680811X13022985131174. PMID 21902942
- [Derived] Tran H, Tran K, Turingan I, Zajkowska M, Lam V, Hawthorne W. Single-incision laparoscopic inguinal herniorraphy with telescopic extraperitoneal dissection: technical aspects and potential benefits. Hernia. 2015 Jun;19(3):407-16. doi: 10.1007/s10029-015-1349-6. Epub 2015 Feb 3. PMID 25644488
- See also: The Sydney Hernia Clinic — http://www.herniaclinic.com.au
- See also: The Sydney Hernia Specialists Clinic — http://www.sydneyherniaspecialists.com.au
- See also: The University of Sydney — http://www.sydney.edu.au/health_sciences/current_students